CLINICAL TRIAL: NCT07236892
Title: Restoring Complex Movement and Locomotion After Paralysis Through Collaborative Copilots: Algorithm Development With Healthy Participants
Brief Title: Towards Restoring Complex Movement After Paralysis: Algorithm Development With Healthy Participants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jonathan Kao, Associate Professor, UCLA ECE & CS, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25-1072; 1DP1HD121548-01 (NIH)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Movement Disorders; Neurorehabilitation; Non-invasive Activity Recording
Keywords: Machine Learning; Algorithm Development
MeSH Terms: conditions — Movement Disorders | interventions — Fixation, Ocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Participants (Experimental): Participants will perform a subset of tasks while non-invasive activity is recorded which may include EEG, EMG, IMUs, fNIRS, eye gaze, or pupillometry.
  Interventions: Behavioral: Participants will perform experimental tasks while undergoing non-invasive activity recordings, which may include EEG, EMG, IMUs, fNIRS, eye gaze, or pupillometry.

INTERVENTIONS:
Behavioral: Participants will perform experimental tasks while undergoing non-invasive activity recordings, which may include EEG, EMG, IMUs, fNIRS, eye gaze, or pupillometry. — Participants may be prompted to imagine, attempt, or perform actions while a task is being performed on a computer, robotic arm, wheelchair, or exoskeleton. Participants may also autonomously perform actions to control each end effector. Participants may be asked to control a cursor to acquire a target or multiple targets. Participants may be asked to pick and place various objects, interact with articulated objects, or perform other motor tasks using a robotic manipulator. Participants may be asked to navigate a wheelchair.

SUMMARY:
Participants will perform experiments with non-invasive activity recordings. The study will record from multiple non-invasive signal sources that reflect motor intent that may include: electroencephalography (EEG), electromyography (EMG), functional near infrared spectroscopy (fNIRS), inertial measurement units (IMUs), eye movements, pupil size, and speech. Participants will wear all or a subset of these sensors and be asked to perform, imagine, or attempt movements or speech. The recorded sensor signals will be decoded to help guide an end effector, which may be a computer, robotic arm, wheelchair, or other assistive device.

These experiments present minimal risk and participants may withdraw participation at any time for any reason. Participants may return for additional experiments if desired and to perform additional comparisons. If a participant withdraws during a comparison, another participant will be recruited to complete collection of data for that comparison.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in the English language

Exclusion Criteria:

* Neurological injury or disease that results in functional paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Normalized Performance | Usually one visit (Day 1), with possible additional study visits usually within a month.
  The normalized performance of the non-invasive assistive interface on a task. Non-invasive signals, which may include electroencephalography, electromyography, functional near infrared spectroscopy, inertial measurements units, eye movements, pupil size, and speech are input into an algorithm that controls an end effector's movements. The end effector, which may be a computer cursor, robotic manipulator, wheelchair, or other assistive device, is used to perform a motor task. The normalized performance is derived from the the performance of the end effector on the motor task, reflecting the overall performance of the non-invasive assistive interface. The minimum value is zero. There is no maximum value, although the values are usually less than 1. Higher is better.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kao, PhD, Principal Investigator — UCLA Neural Engineering and Computation Lab
Locations (1):
- UCLA Neural Engineering and Computation Lab, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
* Identifier data, along with non-invasive activity (e.g., EEG, EMG, fNIRS, IMU, eye gaze) and corresponding behavior (e.g., cursor kinematics, robotic arm joint angles, wheelchair kinematics) will be generated for participants. The species is human, format .bin (binary file), amount per experiment approximately 6 GB.
  * Non-invasive activity and corresponding behavior will be preserved and shared, corresponding to nonidentifiable data collected during experiments.
  * Documentation will be provided to facilitate interpretation of the data.
  * Specialized tools, software, or code are not needed. The data is stored in Python, which is freely available, and can be loaded following documentation.
  * No consensus standard exists. These will be custom datasets for the particular experimental tasks. All data will be de-identified before sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available no later than the time of an associated publication or the end of performance period of the extramural award that generated the data, whichever comes first. DASH, which is an NIH-recommended domain-specific repository, has usually long retention cycles and will often host data "in perpetuity." The PI will not take down the data any sooner.
Access Criteria: Scientific data and metadata will be archived on NICHD Data and Specimen Hub (DASH). DASH automatically assigns a digital object identifier (doi) to data files.
  DASH is an NIH-controlled-access data repository. The NICHD DASH Data Access Committee reviews all requests to access DASH data and biospecimens from identity-verified requesters to determine whether the proposed use is scientifically and ethically appropriate and does not conflict with constraints or research data use limitations identified by the institutions that submitted the research data. The Recipient's institution and the Recipient must sign and agree to the terms and conditions.